CLINICAL TRIAL: NCT02931045
Title: Antiplatelet Therapy Effect on Platelet Extracellular Vesicles in Acute Myocardial Infarction
Brief Title: Antiplatelet Therapy Effect on Extracellular Vesicles in Acute Myocardial Infarction
Acronym: AFFECT EV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Aleksandra Gasecka, Medical Doctor, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: KB/112/2016
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-11

CONDITIONS: Myocardial Infarction
Keywords: extracellular vesicles; inflammation; thrombosis; antiplatelet drugs
MeSH Terms: conditions — Myocardial Infarction; Inflammation; Thrombosis | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ticagrelor (Active Comparator): Ticagrelor: oral, 180 mg once (loading dose) followed by 90 mg twice daily (maintenance dose)
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): Clopidogrel: oral, 300 mg or 600 mg once (loading dose) followed by 75 mg once daily (maintenance dose)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Comparison of ticagrelor with another antiplatelet drug (clopidogrel)
  Other Names: Brilique
  Arms: Ticagrelor
Drug: Clopidogrel — Comparison of clopidogrel with another antiplatelet drug (ticagrelor)
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
Platelet activation and aggregation leads to myocardial infarction. Platelet P2Y12 receptors are essential for platelet activation. Antagonists against the P2Y12 receptor, which are established in secondary prevention of myocardial infarction, have unexplained anti-inflammatory effects. A novel P2Y12 receptor antagonist ticagrelor reduced infection-related mortality compared to clopidogrel, previous standard treatment for patients with myocardial infarction. Activated platelets release pro-inflammatory and procoagulant platelet extracellular vesicles. The investigators assume that decrease in infection-related mortality in patients treated with ticagrelor may be explained by greater inhibition of the release of platelet vesicles by ticagrelor, compared to clopidogrel. This study is expected to identify an additional mechanism of action of ticagrelor, which might contribute to the observed clinical benefits in patients treated with ticagrelor.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Informed consent to participate in the study
* Percutaneous coronary intervention with stent implantation due to first S T elevation myocardial infarction, or first non S T -elevation myocardial infarction
* Administration of a loading dose of clopidogrel

Exclusion Criteria:

* Known coagulopathy
* Known history of bleeding disorder
* Suspicion of intracranial haemorrhage
* Need for oral anticoagulation therapy
* Administration of glycoprotein (GP) II b - III a antagonists
* Cardiogenic shock
* Severe chronic renal failure (estimated glomerular filtration rate < 30 mL/min)
* Severe liver insufficiency
* Chronic dyspnea
* Increased risk of bradycardia
* Autoimmune disease
* Infectious disease
* Neoplasms
* Pregnancy
* Study drug intolerance
* Co-administration of ticagrelor or clopidogrel with strong CYP3A4 inhibitors
* Participation in any previous study with ticagrelor or clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Gasecka, MD, Principal Investigator — 1st Chair and Department of Cardiology, Medical University of Warsaw
Locations (2):
- Laboratory of Experimental Clinical Chemistry, Academic Medical Centre of the University of Amsterdam, Amsterdam, Netherlands
- 1st Chair and Department of Cardiology, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No
The data will be presented in a collective form. If a particular study participant presents with an especially high or low concentration of the studied biomarker , the participant's characteristics may be described separately in a way which does not allow to identify the participant's personal data.

REFERENCES:
- [Background] Gasecka A, Nieuwland R, van der Pol E, Hajji N, Cwiek A, Pluta K, Konwerski M, Filipiak KJ. P2Y12 antagonist ticagrelor inhibits the release of procoagulant extracellular vesicles from activated platelets. Cardiol J. 2019;26(6):782-789. doi: 10.5603/CJ.a2018.0045. Epub 2018 Apr 19. PMID 29671861
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/29398917

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ticagrelor | Clopidogrel
Started | 30 | 30
Completed | 27 | 28
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor | Clopidogrel | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 16 | 35
  >=65 years | 11 | 14 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 22 | 24 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Poland | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Platelet Extracellular Vesicles/ml
Description: Concentration of platelet extracellular vesicles/ml measured with flow cytometry
Time Frame: 6 months following the beginning of antiplatelet therapy
Measure: Median (Inter-Quartile Range); unit: Platelet Extracellular Vesicles/mL
Groups:
- Ticagrelor: Ticagrelor: oral, 180 mg once (loading dose) followed by 90 mg twice daily (maintenance dose)
  27 patients
- Clopidogrel: Clopidogrel: oral, 300 mg or 600 mg once (loading dose) followed by 75 mg once daily (maintenance dose)
  28 patients
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 27 | 28
Platelet Extracellular Vesicles/mL | 2690000 [1460000 to 4190000] | 4310000 [2050000 to 6240000]

2. Secondary Outcome: Concentration of Extracellular Vesicles Exposing Fibrinogen
Description: Concentration of extracellular vesicles exposing fibrinogen/ ml measured with flow cytometry
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Concentration of Extracellular Vesicles Exposing Phosphatidylserine
Description: Concentration of extracellular vesicles exposing phosphatidylserine/ml measured with flow cytometry
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Concentration of Extracellular Vesicles From Endothelial Cells
Description: The concentrations of extracellular vesicles from endothelial cells/ ml measured with flow cytometry
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Concentration of Extracellular Vesicles From Leukocytes
Description: Concentration of extracellular vesicles from leukocytes/ ml measured with flow cytometry
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Ticagrelor: Ticagrelor: oral, 180 mg once (loading dose) followed by 90 mg twice daily (maintenance dose)
  27 patients
  One major bleeding event from the gynecologic tract
- Clopidogrel: Clopidogrel: oral, 300 mg or 600 mg once (loading dose) followed by 75 mg once daily (maintenance dose)
  28 patients
  One major bleeding event from a diabetic foot ulcer
Arm/Group | Ticagrelor | Clopidogrel
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=30) | Clopidogrel (N=30)
One major bleeding event from the gynecologic tract (Reproductive system and breast disorders) | 1 (1) | 1 (1) — In a patient who was eventually diagnosed with endometrial cancer.
One major bleeding event from a diabetic foot ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — In a male patient who had dysregulated diabetes and infection of a diabetic foot.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT02931045/Prot_SAP_000.pdf